CLINICAL TRIAL: NCT02028988
Title: Enzalutamide With External Beam Radiation for Intermediate Risk Prostate Cancer: A Phase II Study
Brief Title: Enzalutamide + External Beam Rt For Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Principal Investigator, Glenn Bubley, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-444
Record Dates: First submitted 2013-12-16; First posted 2014-01-07 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Intermediate Risk Prostate Cancer
Keywords: Intermediate Risk Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzalutamide with External Beam Radiation (Experimental): Enzalutamide
  40 mg orally 4x daily for 6 (28 day +/-3 days) cycles.
  External Beam Radiation Therapy (EBRT) - 7-10 weeks after beginning Enzalutamide
  75.6 to 79.2 Gy in 1.8 Gy fractions for up to 11 weeks.
  *Patients that are unable to complete enzalutamide therapy will still be treated with EBRT
  Interventions: Drug: Enzalutamide; Radiation: External Beam Radiation

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: Xtandi
Radiation: External Beam Radiation

SUMMARY:
This research study is evaluating a drug called enzalutamide in combination with external beam radiation therapy as a possible treatment for prostate cancer. Presently, when participants receive hormonal therapy with radiation therapy for prostate cancer, medications are given to reduce testosterone levels in the blood stream. This leads to side effects such as loss of sex drive, erectile dysfunction (ED) and decrease in muscle strength. The purpose of this study is test another form of hormonal therapy with radiation therapy. The medication called enzalutamide will be used with radiation therapy. Instead of lowering testosterone, enzalutamide blocks testosterone in cells. This study will test if enzalutamide when used with radiation will lower the PSA without causing the side effects associated with medications that lower testosterone in the blood stream.

DETAILED DESCRIPTION:
* The participant will be given a study drug-dosing diary for each of 6 treatment cycles. Each treatment cycle lasts 28 days (4 weeks), during which time the participant will be taking the study drug enzalutamide by mouth (4 pills daily). The diary will also include special instructions for taking the enzalutamide.
* The participant will also be undergoing external beam radiation therapy during the study, for a duration of 8 ½-10 weeks. Treatment will be administered on an outpatient basis. This part of the study is considered standard of care.
* The participant will be required to have fiducial markers placed within the prostate as part of this study. These are very small gold markers that are placed in the prostate. This procedure is similar to the biopsy that the participant had to diagnose their cancer. This procedure is routinely performed to permit imaging and position corrections to improve the precision of the external beam (radiation) delivery (Image Guided Radiation Therapy). The placement of the three gold markers is performed by an Urologist. The fiducials are placed under ultrasound guidance. This is also considered standard of care and is not experimental.
* Planned Follow-up: Participants will be followed on study at a 3 month follow-up after treatment (cessation of enzalutamide). Additional follow-up to assess the status of the participant's cancer will be conducted at the discretion of the treating physicians as part of the participant's routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Study population: Participants must have histologically confirmed malignancy and are candidates for external beam radiation therapy. Patients eligible for this study must have intermediate risk disease defined as PSA values between 10-20 ng/ml and/or T2b-c and/or Gleason grade 7. If all three are present, less than 50% of the core biopsies can be positive.
* Patients previously diagnosed with low risk (Gleason score < 6, clinical stage < T2a, and PSA< 10) prostate cancer undergoing active surveillance who are re-biopsied and found to have intermediate risk disease according to the protocol criteria are eligible for enrollment within 180 days of the repeat biopsy procedure.
* Age 18 years or more.
* Life expectancy of greater than 1 year.
* ECOG performance status ≤ 2 (see Appendix D).
* Participants must have normal organ and marrow function as defined below:
* Leukocytes ≥3,000/mcL
* Platelets ≥80,000/mcL
* Total bilirubin < 2X institutional upper limit
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
* Creatinine < 2x institutional limits .
* The effects of enzalutamide on the developing human fetus are unknown. For this reason and because enzalutamide may be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients must NOT meet any of the following exclusion criteria
* Received an investigational agent within 4 weeks prior to enrollment
* Stage T4 prostate cancer by clinical examination or radiologic evaluation.
* Hypogonadism or severe androgen deficiency as defined by screening serum testosterone less than 50 ng/dL below the normal range for the institution.
* Prior androgen deprivation, chemotherapy, surgery, or radiation for prostate cancer.
* Receiving concurrent androgens, anti-androgens, estrogens, or progestational agents, or received any of these agents within the 6 months prior to enrollment or having taken finasteride or dutasteride within 30 days of registration.
* History of another active malignancy within the previous 5 years other than curatively treated nonmelanomatous skin cancer and superficial bladder cancer. Participants treated for malignancy with no relapse within two years are eligible to participate in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment.
* Unwilling to use contraceptives while on study if relevant to patient.
* History of seizure or any condition or concurrent medication that may predispose to seizure.
* History of loss of consciousness or transient ischemic attack within 12 months prior to enrollment.

  * Clinically significant cardiovascular disease, including:
  * Myocardial infarction within 3 months of enrollment;
  * Uncontrolled angina within 3 months of enrollment;
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within 3 months results in a left ventricular ejection fraction ≥ 45%;
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
  * Hypotension as indicated by systolic blood pressure < 86 mmHg on 2 consecutive measurements at the Screening visit;
  * Bradycardia as indicated by a heart rate < 50 beats per minute at the Screening visit;
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg on 2 consecutive measurements at the screening visit;
  * EKG demonstrating equal to or greater than grade III toxicity according the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
  * History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of oral study drug(s) within 3 months of enrollment.
  * Major surgery within 4 weeks of registration.
  * Previous use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700, TAK-683, TAK-448) or targets the androgen receptor (e.g., enzalutamide, BMS 641988); ketoconazole.
  * Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, places the patient at undue risk, or complicates the interpretation of safety data.
  * Need for any of the medications on the list of drugs to be used with caution or to be avoided (see APPENDIX F).
  * Use of herbal or alternative remedies that may affect hormonal status such as Prostasol or PC-SPES.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bubley, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaplan I, Bubley GJ, Bhatt RS, Taplin ME, Dowling S, Mahoney K, Werner E, Nguyen P. Enzalutamide With Radiation Therapy for Intermediate-Risk Prostate Cancer: A Phase 2 Study. Int J Radiat Oncol Biol Phys. 2021 Aug 1;110(5):1416-1422. doi: 10.1016/j.ijrobp.2021.02.027. Epub 2021 Feb 23. PMID 33636278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from February 2014 to February 2017
Groups:
- Enzalutamide With External Beam Radiation: Enzalutamide
  40 mg orally 4x daily for 6 (28 day +/-3 days) cycles.
  External Beam Radiation Therapy (EBRT) - 7-10 weeks after beginning Enzalutamide
  75.6 to 79.2 Gy in 1.8 Gy fractions for up to 11 weeks.
  *Patients that are unable to complete enzalutamide therapy will still be treated with EBRT
  Enzalutamide
  External Beam Radiation
Period: Overall Study
Arm/Group | Enzalutamide With External Beam Radiation
Started | 64
Evaluable if Treatment Completed | 62
Completed | 62
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 70 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 50
  More than one race | 1
  Unknown or Not Reported | 8
M Stage [Count of Participants; unit: Participants] — Metastatic Stage
  MX: Metastasis cannot be evaluated. M0: The cancer has not metastasized beyond the immediate prostate region. M1: The cancer has metastasized deeper into the body.
  Participants
    MX | 9
    M0 | 50
    M1 | 0
    Unknown | 5
N Stage [Count of Participants; unit: Participants] — Node Stage:
  NX: The regional lymph nodes cannot be evaluated. N0: The cancer has not spread to lymph nodes in the immediate area. N1: The cancer has spread to lymph nodes in the pelvic region.
  Participants
    NX | 12
    N0 | 50
    N1 | 0
    Unknown | 2
T Stage [Count of Participants; unit: Participants] — Tumor Stage:
  T1a: Tumor is found accidentally during a surgical procedure used to treat benign prostatic hyperplasia (BPH). Found in 5 percent or less of the tissue removed.
  T1b: Found accidentally during BPH surgery. Detected in more than 5 percent of the tissue removed.
  T1c: Found during a needle biopsy that was performed because of elevated PSA level.
  T2a: Has invaded one-half (or less) of one side of the prostate. T2b: Has spread to more than one-half of one side of the prostate, but not to both sides.
  T2c: Has invaded both sides of the prostate. T3: Has grown outside the prostate
  Participants
    T1a | 0
    T1b | 0
    T1c | 43
    T2a | 18
    T2b | 1
    T2c | 2
    T3 | 0
Gleason Score [Count of Participants; unit: Participants] — The pathologist looking at the biopsy sample will assign one Gleason grade to the most predominant pattern in your biopsy and a second Gleason grade to the second most predominant pattern. For example: 3 + 4. The two grades will then be added together to determine your Gleason score. Theoretically, Gleason scores range from 2-10. However, since Dr. Gleason's original classification, pathologists almost never assign scores 2-5, and Gleason scores assigned will range from 6 to 10, with 6 being the lowest grade cancer.
  Participants
    6 | 2
    7 | 62
Primary Gleason Score [Count of Participants; unit: Participants] — Because numerous studies suggest that Gleason 3 + 4 tumors (ie, those where pattern 3 is most prevalent but some amount of pattern 4 is also observed) have a better prognosis than Gleason 4 + 3 tumors (ie, those where pattern 4 is more prevalent than pattern 3), contemporary clinical risk prediction now incorporates primary and secondary Gleason pattern.
  Participants
    3 | 38
    4 | 26
Baseline Prostate Specific Antigen (PSA) [Mean (Full Range); unit: ng/mL] | 7.72 [2.96 to 18.50]
Risk Stratification [Count of Participants; unit: Participants] — Men with intermediate-risk prostate cancer are subdivided into favorable and unfavorable subgroups.
  Intermediate risk: Tumor is confined to the prostate, the PSA=10-20, or Gleason Score=7
  Favorable patients were those who had all of the following:
  One intermediate-risk factor (based on the NCCN classification scheme). Gleason Score of 3+4=7 or less. Less than 50% of biopsy cores positive for cancer.
  Those who were classified as unfavorable could have any of the following:
  More than one intermediate-risk factor. Gleason Score of 4+3=7. Greater than 50% positive biopsy cores.
  Participants
    Favorable | 10
    Unfavorable | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PSA at or Below 0.2 ng/ml
Description: Percentage of participants with PSA level of less than or equal to 0.2 ng/ml at the end of six cycles of enzalutamide and EBRT treatment. Post-treatment PSA nadir level has been shown to be a validated intermediate cancer endpoint in similar settings. The chosen cut-off of 0.2 ng/ml was informed by D'Amico et al Lancet Oncology 2012. PSA levels determined through established methods (blood draw and serum analysis).
Time Frame: End of treatment, up to 27 weeks.
Population: Participants who completed treatment are included in this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
percentage of participants
  <=0.2 ng/ml | 79 [69 to 89]
  >0.2 ng/ml | 21 [11 to 31]

2. Secondary Outcome: Median DHEA-S
Description: Median DHEA-S, collected and assessed using established methods. Reference range is 28-640 ug/dL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: The analysis population is comprised of all enrolled patients with evaluable data for this endpoint at each respective timepoint. As treatment went on, some patients dropped out and/or missed appointments and, as such, data was not collected on these patients.
Measure: Median (Full Range); unit: ug/dL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
ug/dL
  Cycle 1: number analyzed (Participants) | 63
  Cycle 1 | 98 [1 to 305]
  Cycle 5: number analyzed (Participants) | 58
  Cycle 5 | 141 [16 to 580]
  End of treatment: number analyzed (Participants) | 57
  End of treatment | 135 [1 to 545]

3. Secondary Outcome: Median Androstenedione
Description: Median androstenedione, collected and assessed using established methods. Reference range is 40-150 ng/dL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
ng/dL
  Cycle 1 | 56.5 [21 to 176]
  Cycle 5: number analyzed (Participants) | 58
  Cycle 5 | 77.5 [18 to 192]
  End of treatment: number analyzed (Participants) | 58
  End of treatment | 76.5 [57 to 215]

4. Secondary Outcome: Median Testosterone
Description: Median testosterone, collected and assessed using established methods. Reference range is 300-1050 ng/dL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
ng/dL
  Cycle 1 | 349.5 [193 to 927]
  Cycle 5: number analyzed (Participants) | 57
  Cycle 5 | 760 [168 to 2330]
  End of treatment: number analyzed (Participants) | 56
  End of treatment | 730.5 [193 to 2760]

5. Secondary Outcome: Median Free Testosterone
Description: Median free testosterone, collected and assessed using established methods. Reference range is 350-1200 ng/dL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
pg/mL
  Cycle 1: number analyzed (Participants) | 63
  Cycle 1 | 66 [10 to 150]
  Cycle 5: number analyzed (Participants) | 58
  Cycle 5 | 100 [24 to 330]
  End of treatment: number analyzed (Participants) | 56
  End of treatment | 86 [10 to 340]

6. Secondary Outcome: Median Estrone
Description: Median estrone, collected and assessed using established methods. Reference range is 12-72 pg/mL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 | 37 [18 to 72]
  Cycle 5: number analyzed (Participants) | 59
  Cycle 5 | 40 [13 to 320]
  End of treatment: number analyzed (Participants) | 58
  End of treatment | 39 [11 to 71]

7. Secondary Outcome: Median Estradiol
Description: Median estradiol, collected and assessed using established methods. The reference range is 13-42 pg/mL for adult males.
Time Frame: Assessed cycle 1, cycle 5, and end of treatment, up to 27 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
pg/mL
  Cycle 1 | 22.5 [5 to 58]
  Cycle 5: number analyzed (Participants) | 57
  Cycle 5 | 45 [13 to 330]
  End of treatment: number analyzed (Participants) | 56
  End of treatment | 45 [10 to 100]

8. Secondary Outcome: Median Bicep Fat Fold Measurement
Description: Median bicep fat fold measurement taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: The analysis population is comprised of all patients who completed treatment with evaluable data for this endpoint at each respective timepoint. As treatment went on, some patients dropped out and/or missed appointments and, as such, data was not collected on these patients.
Measure: Median (Full Range); unit: mm
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
mm
  Baseline | 14 [2.4 to 118]
  End of treatment: number analyzed (Participants) | 55
  End of treatment | 18 [1.2 to 42]

9. Secondary Outcome: Median Tricep Fat Fold Measurement
Description: Median tricep fat fold measurement taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: as for outcome 8
Measure: Median (Full Range); unit: mm
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
mm
  Baseline | 20 [2.8 to 39]
  End of treatment: number analyzed (Participants) | 55
  End of treatment | 24 [1.2 to 42]

10. Secondary Outcome: Median Shoulder Blade Fat Fold Measurement
Description: Median shoulder blade fat fold measurement taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: as for outcome 8
Measure: Median (Full Range); unit: mm
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
mm
  Baseline | 20 [0 to 56]
  End of treatment: number analyzed (Participants) | 55
  End of treatment | 22 [1.2 to 50]

11. Secondary Outcome: Median Waist Fat Fold Measurement
Description: Median waist fat fold measurement taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: as for outcome 8
Measure: Median (Full Range); unit: mm
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
mm
  Baseline | 28 [10 to 58]
  End of treatment: number analyzed (Participants) | 55
  End of treatment | 28 [1.2 to 134]

12. Secondary Outcome: Median Waist Circumference
Description: Median waist circumference taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: as for outcome 8
Measure: Median (Full Range); unit: mm
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
mm
  Baseline | 104.6 [36 to 150]
  End of treatment: number analyzed (Participants) | 55
  End of treatment | 104.6 [12.5 to 134.6]

13. Secondary Outcome: Median Weight
Description: Median weight taken at baseline and end of treatment.
Time Frame: At baseline and end of treatment, up to 27 weeks
Population: as for outcome 8
Measure: Median (Full Range); unit: kg
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 62
kg
  Baseline | 87.35 [64.1 to 138.2]
  End of treatment: number analyzed (Participants) | 58
  End of treatment | 88.26 [61.61 to 142.6]

14. Secondary Outcome: Number of Participants With a Sleep Quality Score of 0 or 1
Description: Sleep quality measure of the Pittsburgh Sleep Quality Index (PSQI) is scored from 0-3 [0=Very bad, 1=Fairly bad, 2=Fairly good, 3=Very good]. The higher the score, the better the sleep quality.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
Participants
  Cycle 1: number analyzed (Participants) | 62
  Cycle 1 | 54
  Cycle 3: number analyzed (Participants) | 58
  Cycle 3 | 43
  Cycle 5: number analyzed (Participants) | 53
  Cycle 5 | 45

15. Secondary Outcome: Urinary Incontinence Median Score
Description: Urinary incontinence evaluated using the Expanded-Prostate Index Composite - 26 (EPIC 26) EPIC-26 evaluates patient's urinary incontinence (4 items). The 4 items are reported on a scale of 0 - 100. A higher score indicates better urinary function.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Median (Full Range); unit: score
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
score
  Cycle 1: number analyzed (Participants) | 61
  Cycle 1 | 100 [52 to 100]
  Cycle 3: number analyzed (Participants) | 57
  Cycle 3 | 100 [43.75 to 100]
  Cycle 5: number analyzed (Participants) | 48
  Cycle 5 | 84.38 [20.75 to 100]

16. Secondary Outcome: Urinary Irritation Median Score
Description: Urinary irritation evaluated using the Expanded-Prostate Index Composite - 26 (EPIC 26). EPIC-26 evaluates urinary irritation/obstruction (4 items). The final score from the 4 items is reported on a scale of 0 - 100. A higher score indicates better urinary function.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Median (Full Range); unit: score
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
score
  Cycle 1: number analyzed (Participants) | 31
  Cycle 1 | 87.50 [43.75 to 93.75]
  Cycle 3: number analyzed (Participants) | 21
  Cycle 3 | 81.25 [62.5 to 93.75]
  Cycle 5: number analyzed (Participants) | 34
  Cycle 5 | 62.5 [12.5 to 93.75]

17. Secondary Outcome: Bowel Function Median Score
Description: Bowel function measure through the Expanded-Prostate Index Composite - 26 (EPIC 26). EPIC-26 evaluates patient's bowel (6 items). The 6 items are reported on a scale of 0 - 100. A higher score indicates better urinary function.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Median (Full Range); unit: score
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
score
  Cycle 1: number analyzed (Participants) | 58
  Cycle 1 | 100 [50 to 100]
  Cycle 3: number analyzed (Participants) | 56
  Cycle 3 | 97.92 [20.83 to 100]
  Cycle 5: number analyzed (Participants) | 52
  Cycle 5 | 89.58 [45.83 to 100]

18. Secondary Outcome: Sexual Function Median Score
Description: Sexual function measure through The Expanded-Prostate Index Composite - 26 (EPIC 26). EPIC-26 evaluates patient's sexual function (5 items). The 5 items are reported on a scale of 0 - 100.A higher score indicates better urinary function.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Median (Full Range); unit: score
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
score
  Cycle 1: number analyzed (Participants) | 58
  Cycle 1 | 62.5 [0 to 100]
  Cycle 3: number analyzed (Participants) | 48
  Cycle 3 | 32 [0 to 100]
  Cycle 5: number analyzed (Participants) | 48
  Cycle 5 | 19.42 [0 to 100]

19. Secondary Outcome: Hormone Function Median Score
Description: Hormone function evaluated by the Expanded-Prostate Index Composite - 26 (EPIC 26). EPIC-26 evaluates patient's hormonal function (5 items). The 5 items are reported on a scale of 0 - 100. A higher score indicates better urinary function.
Time Frame: Measured at cycles 1, 3, and 5.
Population: as for outcome 2
Measure: Median (Full Range); unit: score
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
score
  Cycle 1: number analyzed (Participants) | 60
  Cycle 1 | 97.50 [50 to 100]
  Cycle 3: number analyzed (Participants) | 55
  Cycle 3 | 90 [35 to 100]
  Cycle 5: number analyzed (Participants) | 51
  Cycle 5 | 75 [25 to 100]

20. Secondary Outcome: Number of Participants With a Fatigue Score of 3 or 4
Description: Feeling fatigue measure of the Patient-Reported Outcome Measurement Information System (PROMIS)-Fatigue Short Form is scored from 0-4 [0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much]. The higher the score, the more fatigued the patient is.
Time Frame: Cycles 1, 3, and 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
Participants
  Cycle 1: number analyzed (Participants) | 62
  Cycle 1 | 2
  Cycle 3: number analyzed (Participants) | 57
  Cycle 3 | 13
  Cycle 5: number analyzed (Participants) | 53
  Cycle 5 | 13

21. Secondary Outcome: Median Collagen Type 1 C-Telopeptide
Description: Median Collagen Type 1 C-Telopeptide is a biomarker for bone metabolism measured and analyzed using established methods. Reference range for adult males is 60-1200 pg/mL
Time Frame: Measured at baseline, end of treatment, and at 3 month follow-up, up to 40 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
pg/mL
  Baseline | 295.5 [208 to 379]
  Off-Treatment: number analyzed (Participants) | 58
  Off-Treatment | 397 [310 to 541]
  3 Month Follow-up: number analyzed (Participants) | 57
  3 Month Follow-up | 314 [229 to 407]

22. Secondary Outcome: Median Bone-Specific Alkaline Phosphatase
Description: Median Bone-Specific Alkaline Phosphatase is a biomarker for bone metabolism measured and analyzed using established methods. Reference range for adult males is 7.5-69.8 ug/L
Time Frame: Measured at baseline, end of treatment, and at 3 month follow-up, up to 40 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
ug/L
  Baseline | 11.5 [9.8 to 14]
  Off-Treatment: number analyzed (Participants) | 57
  Off-Treatment | 12 [10.1 to 13.1]
  3 Month Follow-up: number analyzed (Participants) | 56
  3 Month Follow-up | 12.6 [11 to 15.3]

23. Secondary Outcome: Median Procollagen Type II Intact N Terminal Propeptide
Description: Median Procollagen Type II Intact N Terminal Propeptide is a biomarker for bone metabolism measured and analyzed using established methods. Reference range for adult males is 22-87 ug/L
Time Frame: Measured at baseline, end of treatment, and at 3 month follow-up, up to 40 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: ug/L
Arm/Group | Enzalutamide With External Beam Radiation
Number analyzed (Participants) | 64
ug/L
  Baseline: number analyzed (Participants) | 41
  Baseline | 12.8 [10 to 17]
  Off-Treatment: number analyzed (Participants) | 35
  Off-Treatment | 13.5 [11 to 17]
  3 Month Follow-up: number analyzed (Participants) | 33
  3 Month Follow-up | 13.4 [11.2 to 16.6]

ADVERSE EVENTS:
Time Frame: Evaluated while on treatment and up to the 3 month follow up visit, up to 40 weeks.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term. Participants are not being evaluated based on their post-operative treatment option.
Arm/Group | Enzalutamide With External Beam Radiation
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 64/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide With External Beam Radiation (N=64)
Anemia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 11
Cardiac disorders - Other, specify (Cardiac disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Glaucoma (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 9
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal mucositis (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Chills (General disorders) | 3
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 51
Fever (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 3
Abdominal infection (Infections and infestations) | 1
Prostate infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 6
Ejection fraction decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 10
Weight gain (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 5
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 29
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 8
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 2
Sinus pain (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 8
Libido decreased (Psychiatric disorders) | 19
Restlessness (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 5
Urinary frequency (Renal and urinary disorders) | 46
Urinary incontinence (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 6
Urinary tract pain (Renal and urinary disorders) | 13
Urinary urgency (Renal and urinary disorders) | 13
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Breast pain (Reproductive system and breast disorders) | 25
Ejaculation disorder (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 22
Gynecomastia (Reproductive system and breast disorders) | 34
Pelvic pain (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin induration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 13
Hypertension (Vascular disorders) | 40
Hypotension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT02028988/Prot_SAP_000.pdf